CLINICAL TRIAL: NCT04618354
Title: Comparing the Clinical Characteristics of Male Patients With Latent Autoimmune Diabetes ,Classic Type 2 Diabetes and Classic Type 2 Diabetes
Brief Title: Comparing the Clinical Characteristics of Male LADA, T1DM and T2DM Patients
Acronym: LADA
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Other Study IDs: LADA
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Take a blood sample from the patient and extract serum from it for testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LADA group: The patient was diagnosed with late-onset autoimmune diabetes (LADA).
  Interventions: Other: No interventions
- T2DM group: The patient was diagnosed with type 2 diabetes (T2DM).
  Interventions: Other: No interventions
- T1DM group: The patient was diagnosed with type 1 diabetes (T1DM).
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — This clinical study is a retrospective study, and no interventions have been implemented for patients.

SUMMARY:
Diabetes is a common chronic disease in most parts of the world. Diabetes-related complications are harmful to the human body. Different types of diabetes have different levels of harm to the human body. There are also fewer studies on the relationship between specific types of diabetes and clinical diseases such as osteoporosis and Hypogonadism. Therefore, clarifying the differences in the clinical characteristics of adult men with late-onset autoimmune diabetes (LADA) ,Classical type 1 diabetes (T1DM) and type 2 diabetes (T2DM) will help to further understand the effects of diabetes on bone metabolism and sex hormones.

DETAILED DESCRIPTION:
Diabetes is a common chronic disease in most parts of the world. Diabetes-related complications are harmful to the human body. There are also fewer studies on the relationship between specific types of diabetes and clinical diseases such as osteoporosis and Hypogonadism. This study aimed to compare the prevalence of hypogonadism and osteoporosis among male patients with latent autoimmune diabetes (LADA), type 1 diabetes (T1DM) and type 2 diabetes (T2DM) and investigate the protective factors for hypogonadism and osteoporosis in these patients. This cross-sectional study evaluated male patients with LADA, T1DM, and T2DM who visited the endocrinology department of Shanghai Tenth People's Hospital for diabetes management. Sex hormones, lipid profiles, sex hormone-binding globulin (SHBG), glycosylated hemoglobin A1c, beta-cell function, uric acid, and osteocalcin were determined in serum samples. Therefor，clarifying the differences in the clinical characteristics of adult men with LADA, T1DM and T2DM will help to further understand the effects of diabetes on bone metabolism and sex hormones.

ELIGIBILITY:
Inclusion Criteria:

1. 30 ~ 80 years old male;
2. Meet the American Diabetes Association (ADA) definition and standards for diabetes

Exclusion Criteria:

1. having diseases that affect bone and calcium metabolism, such as hyperthyroidism, hyperparathyroidism, hypogonadism, cushing syndrome, rheumatoid arthritis, cirrhosis, or malignant tumor;
2. the use in the past 6 months of drugs that interfere with bone and calcium metabolism, such as sex steroids, vitamin D metabolites, calcitonin, bisphosphonates, and thyroid hormone;
3. moderate or severe liver and renal dysfunction, including serum alanine aminotransferase of 120 IU/L, aspartate aminotransferase of 80 IU/L, and serum creatinine of 120 μmol/L.

4）a history of congenital/hypogonadotropic hypogonadism or hyperthyroidism, or those who received testosterone replacement therapy in the past 6 months were excluded.

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 600 diabetes Patients from Shanghai Tenth People's Hospital were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 632 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Testosterone | 2016-2021
  total testosterone (nmol/L), testosterone (nmol/L) and SHBG (nmol/L). Hypogonadism was defined as total testosterone levels less than 3.0 ng/ml
Bone mineral density | 2016-2021
  Bone mineral density was measured at the lumbar spine, femoral neck, and right hip by dual-energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
HbA1c | 2016-2021
  Glycosylated hemoglobin A1c
FBG | 2016-2021
  patients with fasting blood glucose 6.1mmol/l or more
PBG | 2016-2021
  patients with 2 hour blood glucose 7.8mmol/l or more
FINS | 2016-2021
  metabolic profile fasting insulin (IU/L)
PINS | 2016-2021
  patients with 2 hour blood insulin
TC | 2016-2021
  metabolic profile Total cholesterol (mmol/L)
TG | 2016-2021
  metabolic profile Triglycerides (mmol/L)
HDL-c | 2016-2021
  metabolic profile high-density lipoprotein cholesterol (mmol/L)
LDL-c | 2016-2021
  metabolic profile Low-density lipoprotein cholesterol (mmol/L)
FSH | 2016-2021
  follicle-stimulating hormone
LH | 2016-2021
  luteinizing hormone

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr, Study Chair — Shang hai Tenth People's Hospital, Shanghai, Shanghai, China, 200072
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai M, Cui R, Yang P, Gao J, Cheng X, Sheng C, Li H, Sheng H, Qu S, Zhang M. Incidence and Risk Factors of Hypogonadism in Male Patients With Latent Autoimmune Diabetes and Classic Type 2 Diabetes. Front Endocrinol (Lausanne). 2021 May 31;12:675525. doi: 10.3389/fendo.2021.675525. eCollection 2021. PMID 34135863
- [Background] Zhang M, Sheng C, You H, Cai M, Gao J, Cheng X, Sheng H, Qu S. Comparing the bone mineral density among male patients with latent autoimmune diabetes and classical type 1 and type 2 diabetes, and exploring risk factors for osteoporosis. J Endocrinol Invest. 2021 Aug;44(8):1659-1665. doi: 10.1007/s40618-020-01472-6. Epub 2021 Jan 2. PMID 33387352
- See also: Incidence and Risk Factors of Hypogonadism in Male Patients With Latent Autoimmune Diabetes and Classic Type 2 Diabetes — http://pubmed.ncbi.nlm.nih.gov/34135863/
- See also: Comparing the bone mineral density among male patients with latent autoimmune diabetes and classical type 1 and type 2 diabetes, and exploring risk factors for osteoporosis — http://pubmed.ncbi.nlm.nih.gov/33387352/